CLINICAL TRIAL: NCT00545259
Title: An Open-label, Two-period, Multi-center, Single Dose Study to Assess the Pharmacokinetics of AEB071 in de Novo Liver Transplant Patients
Brief Title: Pharmacokinetic Study of AEB071 in Patients Following Liver Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAEB071B2101
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2008-02

CONDITIONS: de Novo Liver Transplantation
Keywords: Organ transplant, liver, pharmacokinetics, AEB071, immunosuppression
MeSH Terms: interventions — sotrastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AEB071
  Interventions: Drug: AEB071

INTERVENTIONS:
Drug: AEB071

SUMMARY:
The study will evaluate the pharmacokinetic profile of AEB071 in the immediate post-transplant period in patients who have undergone their first liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Primary liver transplant recipients.
* Transplanted liver functioning at an acceptable level by 24 h post-transplant
* Patients started on tacrolimus therapy within 12 h post-transplant

Exclusion Criteria:

* Previous transplantation or multiple organs transplantation
* Acute rejection
* Non-heart beating donor

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
-Pharmacokinetic of AEB071 & its primary metabolite, AEE800 at predose & up to 72 hours post-operatively -Safety & tolerability (vital signs,ECGs,clinical lab evaluations,seroius/adverse events) -AEB071,AEE800 & tacrolimus in blood for both Periods | at predose & 16 timepoints post-dose

SECONDARY OUTCOMES:
-Pharmacokinetics of tacrolimus in presence of AEB071 -Biliary excretion of AEB071 & primary metabolite (AEE800) from patients with a T-tube -Relationship of free drug concentration, α-1 acid glycoprotein concentration & pharmacokinetics AEB071

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (3):
- Novartis investigative site, Berlin, Germany
- Novartis Investigative Site, Padua, Italy
- Novartis investigative site, Zurich, Switzerland

REFERENCES:
- See also: Results from CAEB071B2101 can be found on the Novartis Clinical Trial Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2641